CLINICAL TRIAL: NCT06036225
Title: PREhabilitation for Patients Awaiting a Liver Transplantation: The Development and Feasibility Testing of a Remote Multicomponent pREhabilitation Intervention: PREPARE
Brief Title: PREPARE- Prehabilitation for Patients Awaiting Liver Transplantation: Feasibility and Acceptability Testing.
Acronym: PREPARE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Belfast Health and Social Care Trust (Other)
Collaborators: Queen's University, Belfast (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 21081JB-AS
Record Dates: First submitted 2023-05-03; First posted 2023-09-13 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Liver Transplant
Keywords: Liver transplant; Liver transplantation; Prehabilitation
MeSH Terms: interventions — Preoperative Exercise

STUDY DESIGN:
Intervention Model Description: Focus groups, experience based co-design and a feasibility study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Receiving the prehabilitation intervention (Experimental): All participants will receive the prehabilitation intervention.
  Interventions: Behavioral: Prehabilitation

INTERVENTIONS:
Behavioral: Prehabilitation — Remote prehabilitation multi-component.
  Other Names: Remote prehabilitation

SUMMARY:
This is a study developing a prehabilitation intervention and then testing the acceptability and feasibility of the intervention.

Start date Aug 2022 for Focus groups and Feb 2023 Co-design workshops and feasibility study date pending

DETAILED DESCRIPTION:
This study is using focus groups and experience based co-design workshops to co-design a remote multicomponent prehabilitation intervention for patients awaiting liver transplantation.

Once the intervention is developed it will then be tested for acceptability and feasibility with the liver transplantation cohort in Belfast Northern Ireland.

ELIGIBILITY:
Inclusion Criteria:

* on the transplant waiting list
* grade 3 below for encephalopathy

Exclusion Criteria:

* grade 4 above encephalopathy
* Known adverse reaction to exercise
* New stroke
* lacks capacity to consent

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-07-24 (Actual); Primary Completion 2024-07-24 (Estimated); Study Completion 2024-09-27 (Estimated)

PRIMARY OUTCOMES:
Recruitment | 6 months
  It will be presented in percentage form and will be defined by
  1. Number of participants active on the list.
  2. Number of participants eligible to participate.
  3. Number of participants informed about the iPRehab study.
  4. Number of participants who were interested in participating.
  5. Number of participants recruited.
  6. Number of participants interested but didn't recruit and reasons why.
  7. Number of participants who own a computer/phone/tablet.
  8. Number of participants who can use a computer/phone/tablet independently.
  9. Number of participants who need support to use a device. Detail the support required.
  Min score 0% Max Score 100% Higher values indicate a higher recruitment rate.
Adherence | 6 months
  This will be recorded using percentage and will be defined by
  1. Number of participants who attended 1:1 sessions.
  2. Number of participants who attended the group exercise classes using a class log.
  3. Number of participants who attend the online monthly peer support sessions while active on the liver transplantation waiting list.
  4. Number of participants who accessed the website/web app.
  5. Which sections of the website/web app are utilised and the number of participants who access each section.
  6. Number of participants who wear the activity tracker and report weekly step count.
  Min score 0% Max Score 100% Higher values indicate a higher adherence rate.
Retention | 6 months
  This will be recorded using percentage and will be defined by
  1. Number of participants who completed the baseline assessment.
  2. Number of participants who completed the 12-week iPRehab study.
  3. Number of participants who completed the assessment 1 week post the iPRehab study.
  4. Number of participants who completed the assessment 12 weeks post the iPRehab study.
  5. Number of participants who drop out and the reasons
  Min score 0% Max Score 100% Higher values indicate a higher retention rate.
Acceptability | 6 months
  This will be measured using an acceptability questionnaire.
  Min score 0% Max Score 100% Higher values indicate a higher acceptability.

SECONDARY OUTCOMES:
Physical function | 6 months
  6 minute walk test. This will be recorded in meters covered in the 6 minute duration of the test.
  Min score 0 Max Score 1000
  Higher values indicate better physical function.
Frailty | 6 months
  The Liver frailty index. This index will determine the degree of frailty patients present while awaiting liver transplantation. This scale determines if the patients are frail, pre-frail or robust.
  Min score 1 Max Score 7 Higher values indicate a higher degree of frailty.

CONTACTS AND LOCATIONS:
Overall Officials: Roger McCorry, Dr, Principal Investigator — Belfast HSCT
Locations (1):
- Queen's University Belfast, Belfast, United Kingdom